CLINICAL TRIAL: NCT03899207
Title: Adiyaman University School of Health
Brief Title: Acupressure and Training for Coping With PMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adiyaman University Research Hospital (Other)
Responsible Party: Principal Investigator, Didem Kucukkelepce, Adiyaman Universty, Adiyaman University Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Adiyaman Universty
Record Dates: First submitted 2019-03-20; First posted 2019-04-02 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Premenstrual Syndrome; Acupressure
MeSH Terms: conditions — Premenstrual Syndrome

STUDY DESIGN:
Intervention Model Description: randomize control trail
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- training +acupressure (Experimental): In the training+acupressure group, 10 women were excluded from the study since they could not participate in acupressure application at different times, 2 women were excluded since they had menstrual irregularities and 4 women were excluded since they could not be contacted.
  Interventions: Other: training
- training (Experimental): In the training group, 4 women were excluded since they did not participate in the reminder training, 1 woman was excluded since she had menstrual irregularities, 3 women were excluded since they wanted to withdraw from the study and 3 women were excluded from the study since they could not be contacted.
  Interventions: Other: training +acupressure
- control (No Intervention): In the control group, 4 women were excluded from the study since they could not be reached and 5 women were excluded since they did not agree to participate in the posttest.

INTERVENTIONS:
Other: training +acupressure — .Training+acupressure group; received training for coping with PMS prepared under the guidance of HBM and "The Booklet of Training for Coping with Premenstrual Symptoms" including information about the training given. In addition to the training, acupressure was applied by the researcher twice a week and 24 times in total. Acupressure application was continued with the same frequency until the end of the study (24 times in total for 3 months). One month after the first home visit, reminder training for coping with premenstrual symptoms was given to the women
  Arms: training
Other: training — Training Group; received the training for coping with PMS prepared under the guidance of HBM and "The Booklet of Training for Coping with Premenstrual Symptoms" including information about the training given. One month after the first home visit, reminder training was given to the women.
  Arms: training +acupressure

SUMMARY:
The study was conducted to determine the effect of acupressure and training, given to women under the guidance of health belief model for coping with premenstrual syndrome, on the premenstrual symptoms and quality of life.

This study was conducted to as a randomized controlled trial. The population of the study was composed of all women with PMS registered in FHCs no. 4 and 14 located in the city center. The sample of the study consisted of women including 51 women in training +acupressure group, 55 women in training group and 57 women in control group. The data were collected with Participant Information Form, PMSS and WHOQOL-BREF in the study. Training and acupressure were administered to the acupressure + training group. Only the training for coping with premenstrual syndrome was given to the training group. The data collection forms were reapplied to all groups 12 weeks after the pretest.

DETAILED DESCRIPTION:
Premenstrual Syndrome is an important collection of symptoms affecting approximately one-fifth of women in reproductive age.

Acupressure is an intervention found in the nursing intervention system and defined as applying constant and powerful pressure on certain/specific points of the body in order to reduce pain, provide relaxation and relief, and to prevent or reduce nausea. Many studies conducted in gynecology have shown that acupressure decreased menstrual distress, premenstrual symptoms, back pain in women experiencing dysmenorrhea, labor pain and nausea and vomiting during pregnancy. In addition, it was shown in the studies that training given for PMS decreased the premenstrual symptoms

ELIGIBILITY:
Inclusion Criteria:

Having regular menstruation (between 21-35 days),

not having any psychiatric diagnosis or any gynecological diseases

not using contraceptives,

not having tissue deformity in the extremities.

Exclusion Criteria:

having any psychiatric diagnosis having any gynecological diseases

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2017-06-30 (Actual); Primary Completion 2017-11-20 (Actual); Study Completion 2018-04-20 (Actual)

PRIMARY OUTCOMES:
The Effects of Health Belief Model-Based Training for Coping with Premenstrual Syndrome and Acupressure on Premenstrual Symptoms and Quality of Life | 10 month
  The premenstrual syndrome scale,The lowest score to be taken from the scale is 44 and the highest score is 220. High score shows an increase in the intensity of the symptoms of premenstrual syndrome. If the total scale score is higher than 50% (110) of the highest score (220) in PMS scale, PMS is considered as "present".In the calculation of WHOQOL-BREF scoring, 1st and 2nd items are evaluated independently while the answers obtained from the 3rd, 4th, 26th and 27th questions are reversely scored since they indicate negative statements. The scale does not have a total score. Higher scores obtained from the subscales of the scale indicate that the quality of life level is high.

CONTACTS AND LOCATIONS:
Overall Officials: Didem Simsek Kucukkelepce, phd, Principal Investigator — World Health Organization
Locations (2):
- Turkey (Türkiye) (2):
  - DİDEM, Adıyaman
  - ınönü Universty, Malatya

IPD SHARING:
Plan to Share IPD: No